CLINICAL TRIAL: NCT05729022
Title: Ultrasound-Guided Microendoscopic Versus Fluoroscopic-Guided Lumbar Transforaminal Epidural Steroid Injections: A Randomized Controlled Trial
Brief Title: Ultrasound-Guided Microendoscopic Versus Fluoroscopic-Guided Lumbar Transforaminal Epidural Steroid Injections
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Quantel Medical (Industry)
Responsible Party: Principal Investigator, Marwan Rizk, Principal Investigator, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-2022-0218
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Radiculopathy Lumbar; Disc Disease Lumbar
Keywords: Epidural Injections; Lumbar Manipulation; Fluoroscopy; Ultrasound
MeSH Terms: conditions — Intervertebral disc disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoroscopy (Placebo Comparator): A local anesthetic (2% lidocaine), a 22G, 90mm needle (Quincke spinal needle) is inserted into the skin. Once the needle tip is in its target position, 0.5-5 cc of contrast (Omnipauqe) is injected. If the contrast spread along the spinal nerve into the epidural space, a mixture of 3 cc of 0.125% Marcaine and 40 mg of Depo-Medrol is injected or Diprofos (1/2 ampoule (2 ml) per level).
  Interventions: Radiation: Fluoroscopy
- Ultrasound Microendoscopic (Experimental): A US device with a curvilinear probe and with a microendoscope (EvoTouch+7 Star Scope), inserted into an 18G needle is used. This group will also receive one AP view fluoroscopy (as control) to check for the diffusion of the contrast material in the epidural space.
  Interventions: Device: Ultrasound microendoscopic technique

INTERVENTIONS:
Device: Ultrasound microendoscopic technique — Ultrasound-guided microendoscopic lumbar transforaminal epidural steroid injection
  Arms: Ultrasound Microendoscopic
Radiation: Fluoroscopy — Fluoroscopy-guided lumbar transforaminal epidural steroid injection.
  Arms: Fluoroscopy

SUMMARY:
The purpose of this study is to compare the Microendoscopic combined with ultrasound technique to the standard routinely used X-ray guided transforaminal steroid injection technique.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo screening to determine eligibility. Patients who meet the eligibility criteria will be randomized in a double-blind manner to two groups. Patients assigned to Group A will undergo a fluoroscopy guided procedure while patients in Group B will undergo a microendoscopic combined with ultrasound technique.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 64 years old of either sex
* Disease status of American Society of Anesthesiologists grades I to II
* Patients presenting with single-level disc disease and radiculopathy (L2-L3; L3-L4; L4-L5) for steroid injection
* Confirmation of herniated disk by CT or MRI
* Able to give informed consent

Exclusion Criteria:

* Age under 18 or over 64 years old
* Pregnant women
* Disease status of American Society of Anesthesiologists grades III to IV
* Unable to provide an informed consent
* Radiculopathies at multiple spinal levels
* Non-lumbar herniated discs
* Clinically obvious or known spinal deformity or stenosis
* Previous spine surgery
* Local or systemic infection
* Allergy to steroids, anesthetics, or contrast material
* Uncorrectable coagulopathy and patients on anticoagulation therapy
* Patients who refuse the procedure
* Spine tuberculosis or tumors
* Prior injections within 3 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Intervention success rate | During the procedure.
  The success of the procedure would be indicated by a questionnaire (yes/no answer). This includes the success of visualization under ultrasound and the insertion of the needle within the target position.

SECONDARY OUTCOMES:
Patient satisfaction | 3 weeks after discharge.
  Patient satisfaction towards the procedure is indicated on NRS scale (0-10).
NRS pain score | Before procedure, 30 minutes after the procedure, 1 week and 3 weeks after the procedure.
  Pain score will be assessed on NRS scale from 0-10.
Complications | During procedure.
  Intravascular injection, intraneural injection, subarachnoid injection and patient discomfort.
Procedure time | Beginning of procedure till the end.
  Time taken to complete the procedure.
Ultrasound visibility | During procedure.
  Visualization of the radicular artery and visualization of the nerve root (yes/no answer)

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Rizk, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manchikanti L. Transforaminal lumbar epidural steroid injections. Pain Physician. 2000 Oct;3(4):374-98. PMID 16906179
- [Background] Wu A, March L, Zheng X, Huang J, Wang X, Zhao J, Blyth FM, Smith E, Buchbinder R, Hoy D. Global low back pain prevalence and years lived with disability from 1990 to 2017: estimates from the Global Burden of Disease Study 2017. Ann Transl Med. 2020 Mar;8(6):299. doi: 10.21037/atm.2020.02.175. PMID 32355743
- [Background] Mehta N, Salaria M, Salaria AQ. Comparison of fluoroscopic Guided Transforaminal Epidural Injections of Steroid and Local Anaesthetic with Conservative Management in Patients with Chronic Lumbar Radiculopathies. Anesth Essays Res. 2017 Jan-Mar;11(1):17-22. doi: 10.4103/0259-1162.186868. PMID 28298750
- [Background] Hashemi M, Dadkhah P, Taheri M, Haji Seyed Abootorabi SM, Naderi-Nabi B. Ultrasound-Guided Lumbar Transforaminal Epidural Injections; A Single Center Fluoroscopic Validation Study. Bull Emerg Trauma. 2019 Jul;7(3):251-255. doi: 10.29252/beat-070307. PMID 31392224
- [Background] Jee H, Lee JH, Kim J, Park KD, Lee WY, Park Y. Ultrasound-guided selective nerve root block versus fluoroscopy-guided transforaminal block for the treatment of radicular pain in the lower cervical spine: a randomized, blinded, controlled study. Skeletal Radiol. 2013 Jan;42(1):69-78. doi: 10.1007/s00256-012-1434-1. Epub 2012 May 20. PMID 22609989
- [Background] Engel A, King W, MacVicar J; Standards Division of the International Spine Intervention Society. The effectiveness and risks of fluoroscopically guided cervical transforaminal injections of steroids: a systematic review with comprehensive analysis of the published data. Pain Med. 2014 Mar;15(3):386-402. doi: 10.1111/pme.12304. Epub 2013 Dec 5. PMID 24308846
- [Background] Yang G, Liu J, Ma L, Cai Z, Meng C, Qi S, Zhou H. Ultrasound-guided Versus Fluoroscopy-controlled Lumbar Transforaminal Epidural Injections: A Prospective Randomized Clinical Trial. Clin J Pain. 2016 Feb;32(2):103-8. doi: 10.1097/AJP.0000000000000237. PMID 25803759